CLINICAL TRIAL: NCT04683172
Title: Efficacy Assessment of Transcranial Direct Current STIMulation (tDCS) in Reducing Pain in PALliative Cancer Patients.
Brief Title: Transcranial Direct-current Stimulation (tDCS) Efficacy in Refractory Cancer Pain.
Acronym: STIMPAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STIMPAL; 2020-A2098-31 (Other: ANSM)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cancer Pain; Refractory Pain
MeSH Terms: conditions — Cancer Pain; Pain, Intractable

STUDY DESIGN:
Intervention Model Description: Bicentre, double blinded, randomized, parallel-arm, sham-controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Active tDCS will be delivered daily for 5 consecutive days with the patient either sitting or lying down.A tDCS session generally lasts 20 minutes.
  Interventions: Device: Active Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): Sham tDCS will be delivered daily for 5 consecutive days with the patient either sitting or lying down.A tDCS session generally lasts 20 minutes.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation — tDCS consists of delivering a low-intensity (1 to 2 milliamperes) direct electrical current by means of a pair of electrodes (anode and cathode) applied to the scalp. Electrodes generally have a diameter (round electrode) or a diagonal (rectangular electrodes) ranging from 2 to 3.5 cm.
  To stimulate a given cortical zone, the anode is placed over of the selected zone, generally identified by means of an EEG headset (10/20 System Positioning). For the treatment of pain, the anode is placed over the primary motor cortex (M1) on the contralateral side to the pain or on the left side in patients with diffuse pain. The cathode is placed over a supposedly neutral cortical zone, usually the contralateral supraorbital cortex with respect to the anode. In this study, the stimulation intensity will be 1.5 mA using round sponge electrodes 3.5 cm in diameter.
  Other Names: Active tDCS
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation — The tDCS device has a "Sham" mode that allows for true placebo stimulation. A simulated session is thus designed as a real stimulation session without its effects. Sensations similar to tDCS are created by generating currents only at the start of the session.
  Same modalities as for the Active tDCS procedure will therefore be put in place: a pair of electrodes (anode and cathode) are applied to the scalp.To stimulate a given cortical zone, the anode is placed over of the selected zone, generally identified by means of an EEG headset (10/20 System Positioning). For the treatment of pain, the anode is placed over the primary motor cortex (M1) on the contralateral side to the pain or on the left side in patients with diffuse pain. The cathode is placed over a supposedly neutral cortical zone, usually the contralateral supraorbital cortex with respect to the anode.
  Other Names: Sham tDCS
  Arms: Sham tDCS

SUMMARY:
Pain is a common symptom in palliative care cancer patients and is often insufficiently relieved. The 2010 INCA report showed that France is not an exception to this worldwide observation (synopsis of the 2010 national survey). This report shows that pain is the symptom that these patients fear the most and that it dramatically impacts their quality of life. These patients may experience nociceptive pain related to stimulation of sensory nerve endings by the tumour. When tumour resection is impossible, a symptomatic analgesic treatment is generally proposed, mainly consisting of administration of opioid analgesics. At high doses, this treatment induces adverse effects, especially drowsiness and psychomotor retardation that impair the patient's quality of life.

They may also experience neuropathic pain, secondary to anatomical lesions or functional impairment of nerve structures (peripheral nerves or cerebral or spinal tracts) related to repeated surgical procedures and/or radiotherapy. This type of pain may respond to antiepileptic or antidepressant drugs. At high doses, these treatments also induce adverse effects fairly similar to those observed during treatment of nociceptive pain. As these two types of treatment often need to be coprescribed, these patients frequently present an almost permanent state of drowsiness at the end of life, preventing all normal activities of daily living.

In recent years, noninvasive brain stimulation (NIBS) techniques (transcranial magnetic stimulation (rTMS) or transcranial direct-current stimulation (tDCS)) have been successfully used to treat chronic pain. It was shown that these NIBS techniques can improve pain in cancer patients in the palliative care setting.

DETAILED DESCRIPTION:
tDCS appears to be more suitable than rTMS for the treatment of palliative care patients, who are often difficult to mobilize, as tDCS can be delivered at the patient's bedside and possibly even at home, which is not the case with rTMS. tDCS also appears to be rapidly effective (after 5 sessions) in the context of cancer pain, and this effect lasts longer than that of rTMS.

The proposed treatment of refractory cancer pain by tDCS in palliative care patients is a new treatment modality that is well adapted to hospitalised patients. Each patient will receive 20 minutes of transcranial direct-current stimulation daily for 5 consecutive days.

One arm will receive active stimulation and the control arm will receive sham stimulation. Patients and investigators will be blinded to the type of tDCS.

By improving the patient's activities of daily living, this treatment will enable the patient to return home under good conditions for both the patient and the caregivers. This treatment can also be continued at home. This strategy is consistent with current guidelines in this field, in which the priorities are improvement of quality of life, return home and decreased workload for caregivers.

ELIGIBILITY:
Inclusion criteria

1. Patient with a confirmed cancer at a palliative stage
2. Pain whose mean intensity is greater than or equal to 4/10 in the 48 hours preceding inclusion
3. Pain present on a daily or almost daily basis (at least 4 days out of 7)
4. Pain that has been present for at least 48 hours before inclusion
5. Patients aged 18 or over
6. Patients who can be followed for the duration of the study (i.e. 3 weeks)
7. Patients affiliated to a health insurance plan or entitled
8. Life expectancy estimated at more than 3 weeks
9. Agreeing to participate in the study and having signed an informed consent

Exclusion criteria

1. Inability to self-assess pain and complete self-questionnaires
2. History of head trauma or neurosurgical injury
3. Symptomatic intracranial hypertension (HTIC)
4. Uncontrolled epilepsy
5. Impossibility to correctly positioning the medical device
6. Abuse of drugs or psychoactive substances, at the discretion of the investigator
7. Current major depression or psychosis
8. Pregnant or breastfeeding woman
9. Patient already included in a research protocol on pain
10. Patient under legal protection
11. Absence of affiliation to a social security scheme
12. Specific contraindication to tDCS (intracerebral metal implant)
13. Patients deprived of liberty
14. Patients undergoing psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Mean change in Pain Intensity on the Numerical Rating Scale | Baseline up to Day 8
  Pain intensity will be scored from 0 to 10 (0=No pain, 10 = worst pain) on the Numerical Rating Scale, 3 times daily. Mean variation of the pain NRS between the baseline assessment (Day -3 to Day -1) and the Day 8 assessment will be calculated and compared between arms.

SECONDARY OUTCOMES:
Immediate impact of each tDCS session on pain intensity | Day 0 up to Day 4
  Change in Pain Numerical Rating Scale score measured before and after each tDCS session.
Response rate at the end of treatment | Baseline up to Day 8
  Efficacy of treatment, defined by a ≥ 20% reduction of the mean Numerical Rating Scale score between Baseline and Day 8.
Residual analgesic effect | Baseline up to Day 14
  Pain Numerical Rating Scale scores will be measured 3 times daily. Mean Numerical Rating Scale score will be calculated and compared between arms.
Residual analgesic effect | Baseline up to Day 21
  Pain Numerical Rating Scale scores will be measured 3 times daily. Mean Numerical Rating Scale score will be calculated and compared between arms.
Effects of tDCS on pain | Baseline up to Day 21
  Brief Pain Inventory questionnaire, short form (BPI). Mean variations of scores will be compared between arms.
Effects of tDCS on general symptoms | Baseline up to Day 21
  Edmonton Symptom Assessment System (ESAS). Mean variations of scores will be compared between arms.
Effects of tDCS on anxiety and depression | Baseline up to Day 21
  Hospital Anxiety and Depression Scale (HADS). Mean variations of scores will be compared between arms.
Effects of tDCS on anxiety | Baseline up to Day 21
  (State-Trait Anxiety Inventory (Form Y) (STAI-Y). Mean variations of scores will be compared between arms.
Analgesic treatments consumption | Baseline up to Day 8
  Medication Quantification Scale (MQS). Mean variations of scores will be compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul NGUYEN, MD, Study Director — Clinique Brétéché - Nantes
Locations (2):
- France (2):
  - Clinique Brétéché, Nantes
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No